CLINICAL TRIAL: NCT05847335
Title: The Relationship Between Childhood Traumas, and Personality Beliefs and Emotional Intelligence Abilities in University Students: A Cross-sectional Study
Brief Title: Childhood Traumas, and Personality Beliefs and Emotional Intelligence
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: Sultan Abdulhamid Khan TRH
Record Dates: First submitted 2023-03-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: University Students; Childhood Traumas; Emotional Intelligence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University students' forms: A socio-demographic data form will be given to the participants and the childhood trauma scale, Bar-On emotional intelligence scale and Personality Beliefs scale will be administered.
  Interventions: Behavioral: Survey work

INTERVENTIONS:
Behavioral: Survey work — Childhood Trauma scale, Personality Beliefs questionnaire, Emotional Intelligence scale

SUMMARY:
The aim of this clinical study is to show the effects of childhood traumas on emotional intelligence levels and personality beliefs in university students. The key questions it aims to answer are:

Do childhood traumas have an effect on emotional intelligence levels? Do childhood traumas have an effect on personality beliefs? Do emotional intelligence levels have an effect on personality beliefs? A socio-demographic data form, childhood trauma scale, Bar-On emotional intelligence scale and personality beliefs scale will be administered to the participants.

Researchers will compare Group 1 of those with childhood trauma to Group 2 of those without childhood trauma to see the impact of childhood trauma.

DETAILED DESCRIPTION:
Most of the people are faced with the facts such as more or less stressful factors or some of their wishes are not met during their childhood, and these experiences do not turn into a trauma under normal conditions. However, the severity of the stressful event experienced, the age and self-power of the traumatized individual, and the inconvenience of the family and environmental conditions can turn such experiences into a traumatic process and have psychological consequences that will affect the whole life.

Childhood trauma is defined as the exposure of children to attitudes and behaviors that hinder their physical, emotional, mental or social development and harm their health, by their parents or persons responsible for caring for and educating them, or by strangers. Child neglect and abuse is a health problem that impairs the health and well-being of children and leaves permanent scars throughout their lives.

Although structural biological factors are effective at a certain level in the formation of personality, the character dimension of the personality shaped by psychosocial effects is at least as important as the biological dimension. Among the factors that play a role in the formation of personality disorders, dysfunctional beliefs of the person also play a role. Each personality disorder has its own dysfunctional beliefs. These beliefs are shaped by personality development.

Emotional intelligence is defined as the index of personal, emotional and social competences and skills that will help the individual to cope successfully with the pressure and demands of the environment. In other words, emotional intelligence is the ability of an individual to know himself, to control and motivate himself, to postpone his wishes, to control his emotional changes, to resist obstacles, to approach other people with understanding, to sense their deepest feelings, to establish and maintain effective relationships, and learnable psychological and social skills. . Thanks to these skills, people can maximize their success and satisfaction in life.

Traumatic events experienced in childhood can also affect the personality development of the individual and his emotional reactions to the events he has experienced.

In this study, the significant differences results have been obtained in emotional intelligence levels such as avoidant, dependent-passive-aggressive, antisocial, histrionic, schizoid, paranoid and borderline personality belief levels, and intrapersonal, interpersonal, adaptability, stress management and general mood in those with childhood traumas compared to those without childhood traumas. Moderately reliable results were found between childhood traumas levels, personality beliefs, and emotional intelligence levels. Reliable results could not be obtained between obsessive personality beliefs and emotional intelligence levels.

ELIGIBILITY:
Inclusion Criteria:

1. Those who volunteered to participate in the study,
2. Those who have no problem reading and understanding the semi-structured sociodemographic data form, Childhood Trauma scale, Personality Beliefs questionnaire, and Emotional Intelligence scale,

Exclusion Criteria:

1. Those with any systemic disease,
2. Those who took chronic medication up to two months ago,
3. Those with psychiatric disorders who cannot read and fill the semi-structured sociodemographic data form, Childhood Trauma scale, Personality Beliefs questionnaire, and Emotional Intelligence scale,
4. Those with chronic psychiatric diseases such as schizophrenia,
5. Those with comorbid psychiatric illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-10-14 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Socio-demographic data | Three months
  This was thrived by the researcher to determine the socio-demographic characteristics of the participants (e.g., gender, age, class, region of residence, income status, place of residence, etc.) in accordance with the purpose of the study.

SECONDARY OUTCOMES:
Childhood Trauma Scale | Three months
  Bernstein et al. developed a scale consisting of 28 items, with a total score comprised of five sub-scales measuring sexual, physical, and emotional abuse, and physical and emotional neglect during childhood, as well as combinations thereof. In the original study, Cronbach's alpha values ranged from 0.79 to 0.94. Sar et al. conducted a Turkish validity and reliability study of the scale. In the current study, Cronbach's alpha internal consistency coefficients of the sub-dimensions were found to range between 0.64 and 0.87.

OTHER OUTCOMES:
Personality Beliefs Scale - Short Form (PBQ-SF) | Three months
  The Personality Beliefs Scale was developed by Beck et al. To identify core beliefs about self, other people, and the world, based on cognitive theory and clinical observations, for use in DSM-IV Axis-II personality disorders. Each question in the form addresses avoidant, dependent, passive-aggressive, obsessive-compulsive, antisocial, narcissistic, histrionic, schizoid, and paranoid attitudes and beliefs corresponding to each personality disorder in the DSM, and contains a total of 65 items. Items 64 and 65 were excluded from the assessment of the test. After reading the statements in each item, participants mark how much they agree with them from zero (I do not believe at all) to four (I completely believe). Turkish validity and reliability study was done by Taymur et al. While the total Cronbach reliability coefficient of the scale is 0.92, the reliability coefficients of the subscales range from 0.61 to 0.85.
Emotional Intelligence Scale | Three months
  The emotional intelligence (EI) scale, developed by Bar-On, is a likert-type scale consisting of 87 items. Ratings are as follows: 1: totally agree, 2: agree, 3: undecided, 4: disagree, and 5: strongly disagree. The 88th item on the scale reads "I answered the above statements sincerely and correctly." The questionnaires of those who respond to that statement with "strongly agree" are not taken into consideration. The scale evaluates five sub-dimensions of emotional intelligence: personal skills; interpersonal skills; compatibility; coping with stress; general mood. The Turkish adaptation of the scale was carried out by Acar, and the Cronbach alpha coefficient was found to be 0.92 for the total dimensions of the scale. The low scores obtained from the total scale and its sub-dimensions indicate a high EI.

CONTACTS AND LOCATIONS:
Overall Officials: Özgür MADEN, Principal Investigator — Sultan Abdulhamid Khan Training and Research Hospital
Locations (1):
- Health Sciences University Sultan 2. Abdulhamid Han Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data of the study will be sent when requested by the journal editors and reviewers.
Supporting Information: Study Protocol
Time Frame: At any time
Access Criteria: After contacting the corresponding author, the data will be sent if deemed appropriate.

REFERENCES:
- [Result] Gündüz A, Gündoğmuş İ. The relationship of adverse childhood events on automatic thoughts, intermediate beliefs, schemas, anxiety and depressive symptoms and quality of life in university students. J Clin Psy. 2019;22(1):424-35. DOI: 10.5505/kpd.2019.72621
- [Result] Okan M, Şarlak D. The relationship between childhood treatments, loneliness and fur expression style in young adults. Ege Journal of Medicine. 2022;61(4):530-40. https://doi.org/10.19161/etd.1208937
- [Result] Lobbestael J, Arntz A, Bernstein DP. Disentangling the relationship between different types of childhood maltreatment and personality disorders. J Pers Disord. 2010 Jun;24(3):285-95. doi: 10.1521/pedi.2010.24.3.285. PMID 20545495
- [Result] Cohen LJ, Tanis T, Bhattacharjee R, Nesci C, Halmi W, Galynker I. Are there differential relationships between different types of childhood maltreatment and different types of adult personality pathology? Psychiatry Res. 2014 Jan 30;215(1):192-201. doi: 10.1016/j.psychres.2013.10.036. Epub 2013 Nov 4. PMID 24268580
- [Result] Arıkan A. The Relationship Between Childhood Trauma And Paranoid Personality Disorder Symptoms. CUNY Academic Works. 2016. https://academicworks.cuny.edu/cc_etds_theses/620
- [Result] Bertele N, Talmon A, Gross JJ. Childhood Maltreatment and Narcissism: The Mediating Role of Dissociation. J Interpers Violence. 2022 Jun;37(11-12):NP9525-NP9547. doi: 10.1177/0886260520984404. Epub 2020 Dec 23. PMID 33356780
- [Result] Yalch MM, Ceroni DB, Dehart RM. Influence of Child Abuse and Neglect on Histrionic Personality Pathology. J Trauma Dissociation. 2023 Jan-Feb;24(1):111-124. doi: 10.1080/15299732.2022.2119458. Epub 2022 Sep 2. PMID 36053041
- [Result] Beck AT, Butler AC, Brown GK, Dahlsgaard KK, Newman CF, Beck JS. Dysfunctional beliefs discriminate personality disorders. Behav Res Ther. 2001 Oct;39(10):1213-25. doi: 10.1016/s0005-7967(00)00099-1. PMID 11579990
- [Result] Beck AT, Davis DD, Freeman A. Cognitive therapy of personality disorders. 3rd ed.. New York: Guilford Press; 2015.
- [Result] Fournier JC, Derubeis RJ, Beck AT. Dysfunctional cognitions in personality pathology: the structure and validity of the Personality Belief Questionnaire. Psychol Med. 2012 Apr;42(4):795-805. doi: 10.1017/S0033291711001711. Epub 2011 Sep 13. PMID 21910933
- [Result] Torres A, Garcia-Esteve L, Navarro P, Tarragona MJ, Imaz ML, Gutiérrez F, et. al. P02-397-Personality profile or postraumatic stress disorder? personality characteristics in women victim of chronic intimate partner violence. Eur Psychiatry, 2010;25(S1):1-1. https://doi.org/10.1016/S0924-9338(10)71399-7
- [Result] Kaş AN. An exploration of personality beliefs in women regarding victimaziton of violence in terms of self-compassion and coping strategies. Master's thesis, İstanbul Sabahattin Zaim Üniversitesi, 2021. https://tez.yok.gov.tr/UlusalTezMerkezi/TezGoster?key=v7BkNnnepTnbhn8rNR77LSIEAH-VDUiqPdvLmdGGGb8rMk07tUlfENi2UBkPCCVg
- [Result] Petrides KV, Frederickson N, Furnham A. The role of trait emotional intelligence in academic performance and deviant behavior at school. Pers. Individ. Differ. 2004;36(2):277-93. https://doi.org/10.1016/S0191-8869(03)00084-9.
- [Result] Van der Linden D, Tsaousis I, Petrides KV. Overlap between General Factors of Personality in the Big Five, Giant Three, and trait emotional intelligence. Pers. Individ. Differ, 2012;53(3):175-9. https://doi.org/10.1016/j.paid.2012.03.001.
- [Result] Petrides KV, Mikolajczak M, Mavroveli S, Sanchez-Ruiz MJ, Furnham A, Pérez-González JC. Developments in trait emotional intelligence research. Emot Rev. 2016;8(4):1-7. https://doi.org/10.1177/1754073916650493.
- [Result] Salvador Ferrer CM. How to Influence the New Technologies in the Emotional Intelligence and Communication of Higher Education Student. Emotional Intelligence - New Perspectives and Applications [Internet]. 2012 Feb 1; Available from: http://dx.doi.org/10.5772/31716.
- [Result] Bastian VA, Burns NR, Nettelbeck T. Emotional intelligence predicts life skills, but not as well as personality and cognitive abilities. Pers. Individ. Differ. 2005;39: 1135-45.
- [Result] Delhom I, Satorres E, Melendez JC. Can We Improve Skills in Older Adults? Emotional Intelligence, Life Satisfaction, and Resilience. Psychosoc Interv. 2020;29(3):133-9. http://doi.org/10.5093/pi2020a8
- [Result] Oshri A, Sutton TE, Clay-Warner J, Miller JD. Child maltreatment types and risk behaviors: Associations with attachment style and emotion regulation dimensions. Pers. Individ. Differ 2015;73:127-33. https://doi.org/10.1016/j.paid.2014.09.015.
- [Result] Bernstein DP, Fink L, Handelsman L, Foote J, Lovejoy M, Wenzel K, Sapareto E, Ruggiero J. Initial reliability and validity of a new retrospective measure of child abuse and neglect. Am J Psychiatry. 1994 Aug;151(8):1132-6. doi: 10.1176/ajp.151.8.1132. PMID 8037246
- [Result] Şar V, Öztürk E, İkikardeş E. Validity and Reliability of the Turkish Version of Childhood Trauma Questionnaire. Turkiye Klinikleri J Med Sci. 2012;32:1054-63. doi: 10.5336/medsci.2011-26947
- [Result] Beck AT, Beck JS. The Personality Belief Questionnaire. Unpublished assessment instrument. The Beck Institute for Cognitive Therapy and Research, Bala Cynwyd, Pennsylvania; 1991.
- [Result] Butler AC, Cohen LH, Beck AT. The Personality Belief Questionnaire-Short Form: development and preliminary findings. Cogn Ther Res, 2007;31:357-70.
- [Result] Taymur İ, Türkçapar MH, Örsel S, Sargın E, Akkoyunlu S. Validity and Reliability of the Turkish Version of the Personality Belief Questionnaire- Short Form (PBQ-STF) in the University Students. Klin Psikiyatri Derg. 2011;14:199-209.
- [Result] Bar-On R. Emotional quotient inventory user's manual. Toronto: MHS Inc.; 1997.
- [Result] Acar FT. Duygusal Zekâ Yeteneklerinin Göreve Yönelik ve İnsana Yönelik Liderlik Davranışları ile İlişkisi: Banka Şube Müdürleri Üzerine Bir Alan Araştırması, İstanbul Üniversitesi Sosyal Bilimler Enstitüsü İşletme ve Personel Yönetim-Organizasyon Doktora Programı, Doktora Tezi, İstanbul, 2001.
- [Result] Perry C, Lee R. Childhood trauma and personality disorder. In: Spalletta G, Janiri D, Piras F, Sani G, editors. Childhood Trauma in Mental Disorders: A Comprehensive Approach. Springer Nature; 2020. p.231-55. https://doi.org/https://doi.org/10.1007/978-3-030-49414-8
- [Result] Marusak HA, Martin KR, Etkin A, Thomason ME. Childhood trauma exposure disrupts the automatic regulation of emotional processing. Neuropsychopharmacology. 2015 Mar 13;40(5):1250-8. doi: 10.1038/npp.2014.311. PMID 25413183
- [Result] Back SN, Flechsenhar A, Bertsch K, Zettl M. Childhood Traumatic Experiences and Dimensional Models of Personality Disorder in DSM-5 and ICD-11: Opportunities and Challenges. Curr Psychiatry Rep. 2021 Jul 19;23(9):60. doi: 10.1007/s11920-021-01265-5. PMID 34279729
- [Result] Lafleur DL, Petty C, Mancuso E, McCarthy K, Biederman J, Faro A, Levy HC, Geller DA. Traumatic events and obsessive compulsive disorder in children and adolescents: is there a link? J Anxiety Disord. 2011 May;25(4):513-9. doi: 10.1016/j.janxdis.2010.12.005. Epub 2010 Dec 27. PMID 21295942
- [Result] Schwartz F. Prediction of emotional intelligence and theory of mind in adults who have experienced childhood maltreatment. Unpublished Master's Thesis. Winnipeg, MB: University of Manitoba; 2016.
- [Result] Bozdemir F, Gündüz B. The relationships of attachment styles, parental attidues and traumatic childhood experiences with emotional intelligence. Int. J. Human Sci, 2016;13(1):1797-814. https://www.j-humansciences.com/ojs/index.php/IJHS/article/view/3700
- [Result] Delhom I, Guttierrez M, Mayordomo T, Melendez JC. Does Emotional Intelligence Predict Depressed Mood? A Structural Equation Model with Elderly People. J Happiness Stud. 2018;19:1713-26. https://doi.org/10.1007/s10902-017-9891-9
- [Result] Leible TL, Snell WE. Borderline personality disorder and multiple aspects of emotional intelligence. Pers. Individ. Differ. 2003;37:393-404.
- [Result] Békés V, Beaulieu-Prévost D, Guay S, Belleville G, Marchand A. Trauma-related negative cognitions mediate the relationship between avoidant personality beliefs and impeded response to psychotherapy for PTSD. J. Aggress. Maltreatment Trauma, 2019;28(3):297-312.
- [Result] Krajniak MI, Pievsky M, Eisen AR, McGrath RE. The relationship between personality disorder traits, emotional intelligence, and college adjustment. J Clin Psychol. 2018 Jul;74(7):1160-1173. doi: 10.1002/jclp.22572. Epub 2017 Dec 20. PMID 29266285
- [Result] Perrotta G. Histrionic personality disorder: Definition, clinical profiles, differential diagnosis and therapeutic framework. Arch Community Med Public Health, 2021;7(1):1-5.
- [Result] Reinhard MA, Nenov-Matt T, Padberg F. Loneliness in Personality Disorders. Curr Psychiatry Rep. 2022 Nov;24(11):603-612. doi: 10.1007/s11920-022-01368-7. Epub 2022 Oct 1. PMID 36181573
- [Result] Taylor S, Abramowitz JS, McKay D, Calamari JE, Sookman D, Kyrios M, Wilhelm S, Carmin C. Do dysfunctional beliefs play a role in all types of obsessive-compulsive disorder? J Anxiety Disord. 2006;20(1):85-97. doi: 10.1016/j.janxdis.2004.11.005. Epub 2005 Jan 1. PMID 16325116